CLINICAL TRIAL: NCT03645382
Title: The Effects of Jeju Steaming Onion(Oniro) on Reducing Body Fat of Overweight or Obesity Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Professor, PI, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KO_Oniro_body fat
Record Dates: First submitted 2018-08-16; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Overweight; Diabetes Mellitus; Obesity
Keywords: overweight; body fat; diabetic,; obersity; diabetes mellitus; DM; glycemic
MeSH Terms: conditions — Overweight; Diabetes Mellitus; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- baked barley powder consumption (Placebo Comparator): Subjects randomized to the placebo group received one tablet containing baked barley powder per day (900 mg/day). placebo group consumed one capsules, three times daily before meals, for a total of three capsules consumed per day.
  Interventions: Dietary Supplement: baked barley powder
- jeju steam onion powder consumption (Experimental): Subjects randomized to the test group received one tablet containing jeju steam onion powder per day (900 mg/day). placebo group consumed one capsules, three times daily before meals, for a total of three capsules consumed per day.
  Interventions: Dietary Supplement: jeju steam onion

INTERVENTIONS:
Dietary Supplement: baked barley powder — The baked barley was consumed one capsules, three times daily before meals, for a total of three capsules consumed per day.The baked barley powder capsule had approximately 900 mg/day, 336 mg of baked barley and 564 mg of nondigestible maltodextrin.
  Arms: baked barley powder consumption
Dietary Supplement: jeju steam onion — The jeju steam onion was consumed one capsules, three times daily before meals, for a total of three capsules consumed per day.The jeju steam onion capsule had approximately 900 mg/day, 336 mg of jeju steam onion powder and 564 mg of nondigestible maltodextrin.
  Arms: jeju steam onion powder consumption

SUMMARY:
It is well known that steam onion have benefit effects on controlling the blood sugar, triacylglycerol (TG) and total cholesterol (TC). In this study, the jeju steam onion examined whether it has beneficial effects on reducing body fat of overweight or obesity subjects.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial was conducted to verify the effects of jeju steam onion. Fifty-six healthy male and female subjects aged 20-65 years with normal body weight [25.0 kg/㎡ ≤ body mass index (BMI) < 30.0 kg/㎡] were recruited. The basic framework of the present study was based on a previous study. A 12-week (at each visit; screening, 6-week, 12-week), placebo-controlled, randomized study was conducted with overweight subjects (25.0 kg/㎡ ≤ BMI < 30 kg/㎡). Subjects participants were divided into two group: either Jeju steaming onion or matching placebo (the baked barley powder). Randomization was achieved by computer generated block randomization (placebo : test = 1 : 1).

ELIGIBILITY:
Inclusion Criteria:

overweight(WHO) subjects [25.0 kg/㎡ ≤ body mass index (BMI) < 30 kg/㎡]

Exclusion Criteria:

* uncontrolled blood pressure (blood pressure level more than 140/100mmHg)
* fasting blood sugar level more than 126 mg/dl or taking medications (including blood sugar and anti-diabetic drugs)
* history of serious cardiovascular, pulmonary, gastrointestinal, hepatic, renal and/or haematological disease
* taking a weight change medications within 1 month before study
* participation other obese studies within 2 months before study
* having a known allergy to any ingredient in the investigational product
* participation other intervention studies within 1 months before study
* women who are pregnant or desire to become pregnant during the study period
* having any other medical condition which, in the opinion of the investigator, could interfere with participation in the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline fat mass at 12-week. | at baseline and 12-week follow-up
  The body composition of the study participants was measured via dual-energy X-ray absorptiometry (DEXA) to determine

SECONDARY OUTCOMES:
Change from baseline fat percentage at 12-week. | at baseline and 12-week follow-up
  The body composition of the study participants was measured via dual-energy X-ray absorptiometry (DEXA) to determine
Change from baseline lean body mass at 12-week. | at baseline and 12-week follow-up
  The body composition of the study participants was measured via dual-energy X-ray absorptiometry (DEXA) to determine
Change from baseline whole fat area of L1 and L4 at 12-week. | at baseline and 12-week follow-up
  The abdominal fat distribution was measured at L1 and L4 by computed tomography (CT)
Change from baseline visceral fat area of L1 and L4 at 12-week. | at baseline and 12-week follow-up
  The abdominal fat distribution was measured at L1 and L4 by computed tomography (CT)
Change from baseline subcutaneous fat area of L1 and L4 at 12-week. | at baseline and 12-week follow-up
  The abdominal fat distribution was measured at L1 and L4 by computed tomography (CT)
Change from baseline visceral/subcutaneous fat area ratio of L1 and L4 at 12-week. | at baseline and 12-week follow-up
  The abdominal fat distribution was measured at L1 and L4 by computed tomography (CT)

OTHER OUTCOMES:
Change from baseline weight at 12-week. | at baseline and 12-week follow-up
  Briefly, all data were acquired at baseline and week 12. body weight (kg; Inbody370, Biospace Co., Ltd Korea) was measured.
Change from baseline body mass index at 12-week. | at baseline and 12-week follow-up
  Briefly, all data were acquired at baseline and week 12. BMI was calculated in units of kilogram per square meter (kg/㎡).
Change from baseline height(cm) at 12-week. | at baseline and 12-week follow-up
  Briefly, all data were acquired at baseline and week 12. height(cm) was measured.
Change from baseline waist circumference(cm) at 12-week. | at baseline and 12-week follow-up
  Briefly, all data were acquired at baseline and week 12. waist circumference(cm) was measured.
Change from baseline blood pressure (BP; mmHg) at 12-week. | at baseline and 12-week follow-up
  Briefly, all data were acquired at baseline and week 12. blood pressure (BP; mmHg) was measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Clinical Nutrigenetics/Nutrigenomics, Yonsei University., Seoul, South Korea

REFERENCES:
- [Derived] Jeong S, Chae J, Lee G, Shin G, Kwon YI, Oh JB, Shin DY, Lee JH. Effect of Steamed Onion (ONIRO) Consumption on Body Fat and Metabolic Profiles in Overweight Subjects: A 12-Week Randomized, Double-Blind, Placebo-Controlled Clinical Trial. J Am Coll Nutr. 2020 Mar-Apr;39(3):206-215. doi: 10.1080/07315724.2019.1635052. Epub 2019 Aug 1. PMID 31368861